CLINICAL TRIAL: NCT07100236
Title: Identification of a Novel 29-Gene-Based Subtype of Hepatocellular Carcinoma and Its Correlation With Immunotherapy Efficacy
Brief Title: 29-Gene Liver Cancer Subtype and Immunotherapy Effectiveness
Status: Not yet recruiting | Type: Observational
Sponsor: Junjie Xu (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor-Investigator, Junjie Xu, Associate Chief Physician, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Other Study IDs: 2025-0540
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Primary Hepatocellular Carcinoma
Keywords: Primary Hepatocellular Carcinoma; Immunotherapy; RNA-seq
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novel subtype cohort of HCC
  Interventions: Other: Observational study of 29 - gene - defined HCC subtypes and immunotherapy responsiveness correlation
- Other HCC subtypes cohort
  Interventions: Other: Observational study of 29 - gene - defined HCC subtypes and immunotherapy responsiveness correlation

INTERVENTIONS:
Other: Observational study of 29 - gene - defined HCC subtypes and immunotherapy responsiveness correlation — This is a non - interventional observational study. We will stratify patients with hepatocellular carcinoma (HCC) based on transcriptome sequencing of their tumor samples, specifically using a 29 - gene signature to classify them into different subtypes. Without interfering with patients' existing immunotherapy regimens (which are determined by clinical practice), we will retrospectively collect and analyze data on treatment responses. The goal is to explore the correlation between the 29 - gene - based HCC subtypes and responsiveness to immunotherapy, focusing on differences in outcomes like objective response rate (ORR) and progression - free survival (PFS) across subtypes. This study distinguishes itself by emphasizing observational analysis of pre - existing treatment patterns rather than implementing active interventions, aiming to provide insights into personalized immunotherapy for HCC through genetic subtyping.

SUMMARY:
This clinical study plans to include 350 liver cancer patients from 10 tertiary hospitals nationwide, starting from August 1, 2025, at multiple centers such as the affiliated Run Run Shaw Hospital of Zhejiang University School of Medicine (the leading unit). They will be divided into a new typing queue (100 cases) and another typing queue (250 cases) using the 29 gene set algorithm. The study will collect tumor tissue samples obtained from surgical resection or puncture of patients (meeting the requirements of sample size and tumor cell proportion), perform RNA seq transcriptome sequencing, and extract patient baseline data, clinical pathological characteristics, laboratory test results, treatment information, and follow-up data from the hospital medical record system. The main objective of this study is to observe the disease progression time (TTP) and objective response rate (ORR) of patients after receiving targeted combined immunotherapy. The secondary observations include progression free survival (PFS), overall survival (OS), dynamic changes in tumor markers, liver function status, and survival after progression. The aim is to analyze the correlation between the 29 gene based new subtype of liver cancer and the efficacy of immunotherapy, providing a basis for precise diagnosis and treatment of liver cancer.

DETAILED DESCRIPTION:
This is a multicenter cohort study aimed at exploring the correlation between a novel 29-gene-based subtype of primary hepatocellular carcinoma (HCC) and response to immunotherapy, with the goal of verifying that this new subtype exhibits higher responsiveness to immunotherapy.

Study Population: A total of 350 patients with pathologically confirmed primary HCC will be enrolled from 10 tertiary hospitals across China, with Sir Run Run Shaw Hospital, Zhejiang University School of Medicine as the leading center. Eligibility criteria include: age ≥ 18 years; having measurable tumor lesions per RECIST 1.1; receiving targeted therapy combined with immune checkpoint inhibitors (ICI) after sample collection (with ≥4 weeks interval from prior local treatments if any); availability of qualified tumor samples (≥3g frozen surgical tissues or biopsy specimens sufficient for transcriptome sequencing); and provision of informed consent. Patients will be excluded if they have overlapping local treatments (e.g., TACE, ablation, radiotherapy) during or within 4 weeks of target-ICI combination therapy, concurrent active malignancies (except cured basal cell carcinoma, etc.), severe organ dysfunction (e.g., Child-Pugh Class C liver function, NYHA Class Ⅲ-Ⅳ cardiac function), or other factors interfering with efficacy assessment as judged by investigators.

Study Procedures:

Sample Processing and Subtyping: Tumor samples will undergo RNA sequencing using the Illumina HiSeq platform (outsourced to Hangzhou DIAN Diagnostics company). After quality control, alignment, and quantification, hierarchical clustering based on a 29-gene signature will classify patients into a "novel subtype cohort" (unmatchable to TCGA HCC clusters) and an "other subtypes cohort".

Data Collection: Clinical data will be extracted from electronic medical records, including baseline characteristics (age, gender, Child-Pugh classification), treatment details (target-ICI regimens, doses, cycles), imaging evaluations (enhanced CT/MRI for tumor response assessment per mRECIST), and follow-up data (survival status, tumor marker dynamics).

Outcome Measures:

Primary Outcomes: Time to Progression (TTP, defined as the interval from initiation of target-ICI therapy to first progression per mRECIST) and Objective Response Rate (ORR, proportion of patients achieving complete response [CR, disappearance of arterial enhancement in all target lesions] or partial response [PR, ≥30% reduction in sum of target lesion diameters]). ORR will be assessed at Weeks 8, 16, 24, or progression for each line of therapy; if regimens are changed due to poor efficacy, assessment timelines will be reset for the new regimen, with CR/PR status strictly linked to the corresponding regimen.

Secondary Outcomes: Progression-Free Survival (PFS), Overall Survival (OS), dynamic changes in tumor markers (AFP, PIVKA-II), liver function status at progression, and Post-Progression Survival (PPS).

Statistical Analysis: Group differences will be compared using appropriate tests (t-test, ANOVA, Mann-Whitney U test, Chi-square test, or Fisher's exact test as applicable). Survival analyses (TTP, PFS, OS, PPS) will employ the Kaplan-Meier method with Log-rank tests, and Cox proportional hazards models will evaluate the impact of 29-gene subtyping on progression risk. A p-value < 0.05 will be considered statistically significant.

This study aims to provide evidence for precision immunotherapy in HCC by clarifying the association between the 29-gene-based subtype and immunotherapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Patients who visited multiple centers including Sir Run Run Shaw Hospital, Zhejiang University School of Medicine (the leading center) and were diagnosed with primary hepatocellular carcinoma by surgical pathological histology.
* They received targeted drug combined with immune checkpoint inhibitor treatment after the specimen collection time point (post - surgery or post - puncture) (that is: local treatments such as TACE, ablation, etc. are allowed before the start of targeted - immunotherapy combination treatment, but an interval of ≥4 weeks from the targeted - immunotherapy treatment is required).
* Had measurable tumor lesions at the observation start point (according to RECIST 1.1 criteria), and the tumor response status (including complete response [CR], partial response [PR], stable disease [SD] or progressive disease [PD]) could be judged by imaging examination during the observation (such as post - treatment evaluation).
* Had accessible frozen tumor tissue samples from surgical resection (sample volume ≥3g); or tumor tissue samples obtained by puncture (puncture samples need to meet the pathological diagnosis requirements, and the sample quality can support subsequent transcriptome sequencing and analysis).
* Voluntarily participate in this study and sign the informed consent form. If the subject is unable to read and sign the informed consent form due to incapacity and other reasons, their guardian shall act as the agent for the informed process and sign the informed consent form. If the subject is unable to read the informed consent form (e.g., illiterate subject), a witness shall witness the informed process and sign the informed consent form.

Exclusion Criteria:

* Received any local treatment during the targeted - immunotherapy combination treatment (including during treatment and within 4 weeks after treatment interruption), including:

Transcatheter arterial chemoembolization (TACE), transcatheter arterial embolization (TAE), drug - eluting bead transcatheter arterial chemoembolization (DEB - TACE) and other vascular interventional therapies; Radiofrequency ablation, microwave ablation, cryoablation, laser ablation and other ablation therapies; Stereotactic body radiation therapy (SBRT), three - dimensional conformal radiation therapy, intensity - modulated radiation therapy and other local radiation therapies; Intratumoral injection therapy, high - intensity focused ultrasound (HIFU) and other local physical/chemical therapies.

* Local treatment was initiated before the start of targeted - immunotherapy combination treatment, and the local treatment continued into the targeted - immunotherapy treatment period (that is, there was an overlap between local treatment and targeted - immunotherapy treatment or the interval was < 4 weeks).
* Complicated with other active malignant tumors (except for those with cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma with no recurrence for more than 5 years after surgery).
* Severe impairment of important organ functions:

Liver function: Child - Pugh class C, or total bilirubin > 3×ULN; Renal function: Serum creatinine > 1.5×ULN and estimated glomerular filtration rate (eGFR) < 50ml/min; Cardiac function: New York Heart Association (NYHA) cardiac function class Ⅲ - Ⅳ, or left ventricular ejection fraction (LVEF) < 50%.

* Had uncontrolled active infections, including:

Hepatitis B virus DNA > 2000IU/ml (without receiving antiviral treatment); Hepatitis C virus RNA positive and without receiving antiviral treatment; Active tuberculosis infection, septicemia, etc.

* Had a history of autoimmune diseases and currently still needed to use systemic glucocorticoids (prednisone > 10mg/day) or other immunosuppressive therapies.
* Pregnant or lactating women, or patients planning to become pregnant during the study.
* Had a definite history of allergy to the targeted drugs or immune checkpoint inhibitors involved in the study.
* The researcher believed that there were other factors that might affect the judgment of treatment response (such as uncontrolled hypertension, coagulation dysfunction, simultaneous use of other antineoplastic drugs during targeted - immunotherapy treatment, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with pathologically confirmed primary hepatocellular carcinoma, with accessible tumor samples (surgical/frozen biopsy tissues ≥3g or qualified puncture specimens). They receive targeted-immunotherapy after sample collection, with measurable lesions (RECIST 1.1). Local treatments are allowed if not overlapping with target-immunotherapy (interval ≥4 weeks). Excluded: active malignancies/organ dysfunction/uncontrolled infections/autoimmune diseases/pregnancy. All provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Disease Progression Time (TTP) | From target-ICI therapy start, assessed at baseline, Week 8, 16, 24, progression/termination. Max 24 months through study end. Data for all time points.
  Time from initiation of target-ICI therapy to first documentation of disease progression per mRECIST criteria. Progression includes:
  Target lesions: ≥20% increase in sum of arterial-enhancing diameters (vs baseline) + absolute increase ≥5mm; Non-target lesions: New lesions or definite progression of existing non-target lesions; Distant metastasis: New lung, bone, or lymph node metastases.
Objective Response Rate (ORR) | From target-ICI therapy start, per regimen: Week 8, 16, 24, progression/termination. New regimens: same time points (reset). Max 24 months through study end. Data for all.
  Proportion of patients achieving Complete Response (CR: disappearance of arterial enhancement in all target lesions) or Partial Response (PR: ≥30% reduction in sum of target lesion diameters).

SECONDARY OUTCOMES:
Progression - Free Survival (PFS) | From target-ICI therapy start, assessed via imaging (baseline, every 8 weeks) and survival follow-up. Max 24 months through study end. Data for all time points.
  Time from target-ICI therapy start to first disease progression (per mRECIST) or any-cause death (whichever occurs first).
Overall Survival (OS) | From target-ICI therapy start, assessed via regular follow-up. Max 24 months through study end. Survival curves; data for all time points.
  Time from target-ICI therapy start to any-cause death; lost-to-follow-up patients censored at last follow-up.
Alpha-FetoProtein (AFP) | From target-ICI therapy start, assessed at baseline, every 4 weeks. Max 24 months. Data for all time points.
  Monitoring of alpha-fetoprotein (AFP) for ≥20% increase (vs baseline) lasting ≥4 weeks, combined with imaging to predict progression risk.
Protein Induced by Vitamin K Absence or Antagonist II (PIVKA-II) | From target-ICI therapy start, assessed at baseline, every 4 weeks. Max 24 months. Data for all time points.
  Monitoring of protein induced by vitamin K absence/antagonist-II (PIVKA-II) for ≥20% increase (vs baseline) lasting ≥4 weeks, combined with imaging to predict progression risk.
Child-Pugh Class | From target-ICI therapy start, synchronized with progression. Included in 24-month data.
  At disease progression, collect Child-Pugh class data. Compare with baseline (excluding drug-induced liver injury) to analyze direct impact of tumor progression on liver function impairment.
Total Bilirubin | From target-ICI therapy start, synchronized with progression. Included in 24-month data.
  At disease progression, collect total bilirubin data. Compare with baseline (excluding drug-induced liver injury) to analyze direct impact of tumor progression on liver function impairment.
Albumin | From target-ICI therapy start, synchronized with progression. Included in 24-month data.
  At disease progression, collect albumin data. Compare with baseline (excluding drug-induced liver injury) to analyze direct impact of tumor progression on liver function impairment.
Internationalnormalizedratio (INR) | From target-ICI therapy start, synchronized with progression. Included in 24-month data.
  At disease progression, collect INR (International Normalized Ratio) data. Compare with baseline (excluding drug-induced liver injury) to analyze direct impact of tumor progression on liver function impairment.
Post-Progression Survival (PPS) | From disease progression (post target-ICI start), follow-up post-progression. Max 24 months post-progression through study end. Data for all time points.
  Time from disease progression to death or study end. Record post-progression treatments (targeted drug change, local therapy) and analyze impact on survival.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences, Chaoyang, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat - sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Affiliated Hospital of Naval Medical University (Shanghai Eastern Hepatobiliary Surgery Hospital), Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-07-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT07100236/Prot_ICF_000.pdf